CLINICAL TRIAL: NCT03599102
Title: Enhancing Kidney Donation Through Live Organ Video Educated Donors (LOVED) Study Phase
Acronym: LOVED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Pro00031456
Record Dates: First submitted 2016-12-01; First posted 2018-07-26 (Actual); Last update posted 2021-05-18 (Actual); Status verified 2021-05

CONDITIONS: Kidney Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LOVED intervention (Experimental): Intervention group receives the LOVED program, an 8-week program where participants receive video education modules, and weekly video chat sessions with other end-stage renal disease patients and a prior living kidney African American recipient. The program aims to increase knowledge and skills on how to promote individual strategies on how to ask for a kidney from others.
  Interventions: Behavioral: LOVED Intervention
- Standard Care (No Intervention): Standard interaction with transplant center and physician care.

INTERVENTIONS:
Behavioral: LOVED Intervention
  Arms: LOVED intervention

SUMMARY:
LOVED stands for the Living Organ Video Educated Donors (LOVED) program. It is a culturally tailored program for African Americans to reduce the disparity of low rates of living kidney donation. It is a mobile health delivered platform that does not require transplant center visits, thus increasing the reach of the program compared to center-based program to enhance living kidney donation. The purpose of LOVED is to give education and encouragement to those who need a kidney transplant and teach about the process of living donation to be better educated when approaching others about donating a kidney. The ultimate goal of the program is to increase the number of living kidney donor transplants, especially among African Americans in South Carolina. The program was created to educate those in need of a kidney about the donor process, to dispel myths about living donation, discuss who can be asked to donate and develop and practice skills to start asking others for a living kidney donation. The program is designed to be completed using a tablet computer and is made up of weekly video education clips, resources, short quizzes to reinforce the learning points and weekly video chat sessions with others who need a kidney led by a "navigator" who was once a living donor kidney recipient. The video clips are made up of stories and brief educational messages from transplant center staff, physicians, former donors and recipients. The video chat sessions were designed to solve and address individual issues for those enrolled in the program and to give a sense of community as they continue on their journey to find a kidney. This randomized control trial uses groups of 6-9 participants in each LOVED group that lasts 8-weeks each. A total of 60 participants will be recruited with 30 assigned to LOVED and 30 assigned to a standard care groups. This program is funded by a grant from the National Institute of Health and was developed at the Medical University of South Carolina.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years old
* African American
* Legally competent
* Able to read and speak in English
* Able to use tablet computers (after instruction)
* Able to use cell phone
* 5 years or less on the kidney waitlist with active status including pre-emptive and ESRD patients on dialysis
* 10 years or less on dialysis

Exclusion Criteria:

* Patients who have currently identified PDs moving through the evaluation stage

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-04 (Actual); Study Completion 2018-02 (Actual)

PRIMARY OUTCOMES:
Participant adherence to study protocols | Assessed at 8 weeks
  Tolerability as defined by % retention to study (% of participants who self-remove from the study) Fidelity as defined by %adherence to chat sessions and completion %of video modules.
Change in knowledge about living donation | Change between 0 and 8 weeks and change between 0 and 6 months
  Score measures for self-efficacy, knowledge and attitudes to approach others to be a living donor
  -LDKT Knowledge Scale (knowledge) (15 item T/F); each correct response adds 1 point. 0-15 range with higher numbers represent higher knowledge.
Change in attitudes on living donation | Change between 0 and 8 weeks and change between 0 and 6 months
  LDKT Concerns Scale (i.e., measuring attitudes) (21 T/F with one point for each statement suggestive of more worry); 0-21 range with higher results representing more concerns about LDKT.
Change in self-efficacy to ask others to be a living donor | Change between 0 and 8 weeks and change between 0 and 6 months
  Willingness to Discuss LDKT Scale (i.e., measuring self-efficacy (SE)) (1 item each for family, friends, and strangers7 pt. Likert scale) 1-7 range with higher values representing higher SE to approach others about living donation

SECONDARY OUTCOMES:
Completing living donor kidney transplantation | 8 weeks, 6 months
  % who identify potential donors, % elected to be screened and, % completing Living donor kidney transplantation (from clinical records compared between groups)

OTHER OUTCOMES:
Assessment of making autonomous decisions | 8 weeks
  Shared Decision Making Questionnaire (SDM-Q-9), a 6 question 4-item Likert scale (1=strongly agree to 4=strongly disagree) involved decision making between the participant and Loved Navigator. Questions were averaged (range 1-4). Lower scores represent better ability to make decisions.
Assessment of feelings of trust | 8 weeks
  Assess if the participant feels distrust of study staff, and medical providers during after the trial. Abbreviated Trust Measure, 3 question, 4-item Likert scale between participant and navigator. Question scores were averaged where higher scores indicated more trust (range 1-4).
Assessment of cultural competency | 8 weeks
  Assess feelings of inclusion based on race during study process. Experiences of Discrimination, a 5 question, 4-tem Likert scale. Questions were averaged (range 1-4). Higher sum scores represent higher trust perceptions.
Assessment of communication satisfaction | 8 weeks
  Assess feelings of how the communication was administrated during the study. Communication Effectiveness Questionnaire, a 9 question 5-item Likert scale between the participant and the navigator, research staff and renal transplant team. Questions were averaged (range 1-4). Higher sum scores represent higher communication perceptions.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Treiber, PhD, Principal Investigator — Medical University of South Carolina; Baliga Baliga, MD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No